CLINICAL TRIAL: NCT02325869
Title: DebriS Interventional REmoval in ACS (DESIRE-ACS) Study to Assess the Safety and Performance of the ECA Bell Balloon in Subjects Undergoing Coronary Percutaneous Interventions.
Brief Title: Clinical Study Protocol - Debris Interventional Removal in ACS (DESIRE-ACS)
Acronym: DESIRE-ACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Angioslide Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0013.CTIL
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Disease; Acute Coronary Syndrome; Coronary Occlusion
Keywords: Acute Coronary Syndrome, Coronary Occlusion, catheter
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome; Coronary Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bell Balloon Catheter (Experimental): The Bell Balloon Catheter is designed to help the physician capture some of this material that may have broken off.
  Interventions: Device: Bell Balloon Catheter

INTERVENTIONS:
Device: Bell Balloon Catheter — An angioplasty procedure to open the blockage in blood vessels will be performed. Standard angioplasty procedure includes local analgesia of the groin area and a small cut through which the procedure will be performed. An introducer sheath (thin tube) will be inserted. The Bell Balloon dilatation will then be inserted. The Bell Balloon works in fashion similar to standard balloon with the same physical and behavioral characteristics. Upon deflation, debris from the blockage is withdrawn into the cavity formed between the deflated balloon and its outer capsule. Then balloon is retracted and retrieved through the guiding catheter, together with the captured debris and trap it between the outer surface of the balloon and the inner surface of the membrane.

SUMMARY:
DebriS Interventional REmoval in ACS (DESIRE-ACS) Study to assess the safety and performance of the ECA Bell balloon in subjects undergoing coronary percutaneous interventions.

DETAILED DESCRIPTION:
Coronary arterial disease (CAD) is defined as obstruction of blood flow into the coronary arteries (i.e. the arteries that supply blood to the heart muscle). Patients with symptoms of coronary artery disease usually suffer from stable angina pectoris (chest pain or discomfort), unstable angina pectoris, or a myocardial infarction (heart attack). The symptoms range from mild angina, to moderate or severe angina.

In some cases of CAD the blood vessel is chronically totally blocked (total occlusion), stopping blood flow through the blocked blood vessel. In these cases a minimally invasive treatment or a surgery may be needed. "Minimally invasive procedures" consist of angioplasty or stent placement. The procedure is performed under local anesthetic with the patient lying on their back.

Angioplasty is a routine, well known, non-surgical procedure that is performed by making a small incision of the skin in the groin through which a catheter (narrow tube) and a guidewire (a thin metal wire) are inserted to reach the blocked artery. After reaching the blocked artery and crossing the blockage with a guidewire, a tiny balloon is inflated inside the artery to open the blockage. During the course of this procedure small pieces of the material that is causing the blockage may break off and be carried by the blood stream to other parts of the body where they may lodge and cause damage by blocking the blood flow . The Bell Balloon Catheter is designed to help the physician capture some of this material that may have broken off.

ELIGIBILITY:
Inclusion Criteria:

Clinical criteria

1. Subject is ≥18 years of age.
2. Subject with acute coronary syndrome (STEMI or NSTEMI).
3. Candidate for percutaneous coronary intervention (PCI) in native coronary artery.
4. Anticipated patient life expectancy of at least 1 year since enrollment.
5. Subject is male or a non-pregnant female.
6. Subject has provided written informed consent.
7. Subject is able and willing to adhere to the required follow-up visits and testing.

Angiographic Criteria

1. Lesions amendable to PCI.
2. Angiographically thrombotic-appearing lesion that amenable to PCI.
3. Lesion(s) is located within the native vessel and has ≥ 50% but <100% stenosis.
4. The target lesion should be at least 10mm proximal to the proximal edge of a stented lesion.
5. Only a single lesion will be treated by the investigational device.
6. Vessel has thrombolysis in myocardial infarction (TIMI) grade 1 or higher flow before the use of the investigational device.
7. Reference vessel diameter, where the Bell balloon is to be placed, is 3-4mm in diameter by angiographic visual estimation.

Exclusion Criteria:

Clinical Criteria

1. Women except those whose menstrual periods have not occurred for more than one year after menopause or those who have had sterilization surgery (tubal ligation) or hysterectomy
2. Known contraindication to the use of heparin or bivalirum (Angiomax).
3. Known contraindication to the use of dual anti-platelet therapy
4. Known hypersensitivity to contrast media which cannot be adequately pretreated.
5. Subject has renal insufficiency, defined as baseline creatinine level ≥ 2.0 mg/dl.
6. Subject has a known history of neutropenia (WBC <3,000/mm3) or significant anemia.
7. Subjects has a known history of coagulopathy or thrombophilia [prothrombin International Normalized Ratio (INR)>1.5, Platelet count<80,000/ μL], that has not resolved or has required treatment in the past 6 months.
8. Major bleeding within 6 months of index procedure.
9. A planned invasive surgical procedure within 30 days.
10. Undergone cardiac surgery within the past 30 days or has a planned surgical procedure within 30 days from study procedure
11. Left ventricular ejection fraction < 25%
12. The patient is in cardiogenic shock or hemodynamic unstable
13. Cerebrovascular Accident (CVA) or TIA within the past 6 months.
14. Exclusions that preclude placement of the bell balloon per the Instruction for Use
15. Subject not capable of understanding and signing the Informed Consent form.

Angiographic Criteria

1. Anatomical exclusions that preclude placement of the bell balloon per the Instruction for Use.
2. Target lesion inside or within 10mm of a prior stent
3. Target lesion distal to a prior placed stent
4. Severe calcification at the lesion site or proximal to it.
5. Aorto-ostial lesions
6. Bifurcation lesions (side branch diameter ≥ 2.0mm)
7. Severe coronary artery tortuosity (Angulation >450)
8. Target lesion is totally occluded, or Thrombolysis in Acute MI (TIMI flow 0) despite pre-dilatation with small caliber balloon
9. Coronary artery spasm in the absence of a significant stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The rate of major adverse cardiac events (MACE) | Up to 30 (+/-7) days post procedure
  Defined as a composite of cardiac death, all myocardial infarction (Q wave and non-Q wave), and target lesion revascularization (PCI and CABG)
Angiographic and Device Success | During procedure and up to 30 (+/-7) days post procedure
  Defined as patent vessel with stenosis <50% with a final TIMI flow grade 3 (visually assessed by angiography) without side branch loss, flow-limiting dissection, or angiographic thrombus and embolic material retrieval.
  * Thrombolysis In Myocardial Infarction (TIMI) flow grade at the end of the revascularization procedure, compared to baseline.
  * ST resolution level in patients with ST-Elevation Myocardial Infarction (STEMI).
  * Myocardial Blush Grade (MBG) at the end of procedure, compared to baseline
Performance - Device success | During procedure and up to 30 (+/-7) days post procedure
  Defined as ability to deliver, deploy, and intact retract retrieval of the study device and retrieve embolic material

CONTACTS AND LOCATIONS:
Overall Officials: Giora Weisz, Prof. M.D, Principal Investigator — Chairman, Department of Cardiology. Shaare Zedek Medical Center, Jerusalem Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel